CLINICAL TRIAL: NCT03809403
Title: Influence of the Surgical Technique Used for Colectomies on the Concentration of Circulating Tumor DNA and the Presence of Circulating Tumor Cells: Comparison of the "no Touch" Technic With Either First Clamping of the Mesenteric Vessels or First Mobilization of the Tumor Followed by Clamping.
Acronym: ADNCHIR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: APHP180453
Record Dates: First submitted 2018-12-20; First posted 2019-01-18 (Actual); Last update posted 2019-03-14 (Actual); Status verified 2019-02

CONDITIONS: Colorectal Cancer
Keywords: Colorectal cancer; Surgical Technic; No touch technic; Circulating Tumor DNA; Circulating Tumor Cells
MeSH Terms: conditions — Colorectal Neoplasms; Neoplastic Cells, Circulating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 2 samples of 6ml of peripherical blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- "No touch" group:: Patients with left sided colic adenocarcinoma who underwent left colectomy with an early ligation of mesenteric vessels
- "Mobilisation first" group: patients with right colic adenocarcinoma who underwent right colectomy with early mobilisation of the tumor followed by the ligation of the vessels.

SUMMARY:
Colectomy is the most commonly used therapeutic approach for the treatment of non-metastatic colorectal cancer. This approach is generally very effective however the rate of recurrence and the appearance of metachronous metastasis remains a major problem in the postoperative period. One of the hypothesis that can explain this tumor progression is the dissemination of tumor cells at the time of tumor mobilization. In this work, we wish to verify this hypothesis by comparing two surgical technics used in our department for left or right colectomies: respectively either first section of the mesenteric vessels followed by the mobilization of the tumor or first mobilization of the tumor followed by the section of the mesenteric vessels. To evaluate the dissemination, we will study two disseminations markers that have shown their prognostic value: i) circulating tumor cells (which represent a direct marker of dissemination) and ii) tumor circulating DNA (which is an indirect marker) but has the advantage of being more representative of all tumor clones and therefore the tumor burden released into the blood at the time of surgery).

DETAILED DESCRIPTION:
A / Epidemiology of colorectal cancer

Colorectal cancer remains the third most common cancer in France in 2017 with an incidence of about 44,000 new cases in 2017 and nearly 18,000 deaths each year. The ColoRectal Cancer (CRC) ranks second among cancer deaths behind lung cancer and breast cancer. Thanks to diagnostic and therapeutic progress, the mortality rate decrease of 1.5% in men and 1.1% in women between 2005 and 2012.

Despite these numbers, colorectal cancer has a good prognosis when diagnosed at an early stage. In fact, the 5-year relative survival is 91% for localized stages (stage I and II) and 70% for stages with locoregional and lymph nodes invasion (stage III). On the other hand, about 25% of the patients at the time of diagnosis have metastasis (stage IV), with a survival at 5 years of 11%. Those data explain that the mortality of this cancer is mainly due to the spread of the primary tumor to secondary locations, mainly liver or lung.

The unstable microsatellite phenotype (ISM) is an important colonic carcinogenesis pathway, find in approximately 15% of operable colorectal cancers (CRC) and may be of sporadic or hereditary origin. Several studies have shown that patients with MSI tumors have a better prognosis than patients with stable microsatellite tumors (SSM) due to a better response to platinum-based chemotherapy. The determination of this status therefore determines the adjuvant treatment of CRC and is determined in anatomopathology on the analysis of the operative specimen.

B / The place of surgery in the care of the CCR:

Currently, the (tumor node metastasis (TNM) classification is used to establish therapeutic management. Stages I are treated by surgery alone. Stages II are treated by surgery alone in the absence of risk factors for recurrence and with adjuvant chemotherapy if not. Stages III are treated by surgery and adjuvant chemotherapy within 8 weeks and for 6 months. For the stages IV (metastatic), the management of those patients is discussed on a case-by-case basis according to the symptomatic or non-symptomatic nature of the primary tumor and the resectability or non-resectability of the metastasis. If there is no contraindication, most of these patients are treated with first-line chemotherapy, then reassessed every 2 to 3 months.

C / Surgical technic:

Surgical treatment depends on tumor localisation:

In the case of a tumor located on the right colon, from the caecum to the middle of the transverse colon, a right colectomy is performed associated with lymph node dissection along the superior mesenteric vessels.

In the case of a tumor located on the left colon, from the middle of the transverse colon to the rectum, a left colectomy is performed with a dissection centered on the inferior mesenteric artery.

In current practice, there are different surgical technics for both types of left and right colectomies. One of the main differences between those technics is the section of vessels (superior or inferior mesenteric vessels):

The so-called "no touch" technic involves a ligation of the mesenteric vessels before any tumor mobilization. This technic is the one used systematically at Saint Antoine Hospital for left colectomy because of the easy dissection of the inferior mesenteric artery and vein in the absence of mobilization of the left colon, those vessels being at a distance from other elements (the left ureter is visualized before the ligation of the inferior mesenteric artery).

An other technic is to first mobilize the tumor to have an optimal exposure of the vessels before the ligation. This technic is the one routinely performed at Saint Antoine Hospital for the right colectomies because of the anatomy of the ileocolic artery and the right colic artery at the origin of which is performed the lymphadenectomy. Indeed the complete mobilization of the right colon allows a section of the adhesions between the right mesocolon (which contains the colonic vessels) and the duodenum and the right ureter. In this way, the section of the right colic vessels can be made at the origin with good control of adjacent structures. Moreover, the lymph node dissection is systematically performed by laparotomy: indeed even for colectomies performed under laparoscopy it is necessary to make a mini-laparotomy incision in order to extract the operative piece and to perform the anastomosis.

Currently, no difference has been demonstrated in terms of survival without recurrence and overall survival between those different technics.

Moreover, the choice of the approach, laparoscopic or by laparotomy, depends on the comorbidities of the patient, severe respiratory failure may be a contraindication to laparotomy and its history: one or more previous surgeries by laparotomy is considered as a contraindication to laparoscopy.

D / Circulating tumor DNA (ctDNA) and Circulating Tumor Cells (CTC) in colorectal cancer:

One of the metastatic extension factors of colorectal tumors treated at a localized stage (stage II and III) is the dissemination of circulating tumor DNA and circulating tumor cells in the peripheral blood.

Tumor cells witch migrate into the blood and lymphatic vessels from a tumor (primary or metastasis) are called circulating tumor cells (CTCs). Some of these have a tumor inducing potential (responsible for relapses) or the ability to form metastasis with time.

Advances in molecular biology technologies (high-throughput sequencing and digital polymerase chain reaction (PCR), for example) have made possible to consider the exploration of circulating tumor DNA, which is present in small quantities in plasma. The amount of ctDNA is proportional to the tumor burden. Thus the mutations of the tumor's DNA (or somatic mutations) can be identified from the ctDNA, the mutations having a theranostic impact on the KRAS, NRAS and BRAF genes could be identified in the ctDNA of patients presenting colorectal cancers. These mutations can thus serve as tracers, the amount of tumor DNA can also be monitored and DNA methylation tests can also be specific for the tumor DNA. The presence of these molecular abnormalities can therefore be used to detect CTCs and ctDNA in these patients. Several studies, initially conducted in the context of breast cancer,have shown the interest of these two parameters in the monitoring and follow-up of patients with CRC: indeed their short half-life of a few minutes to a few hours allows a follow-up in real time their kinetics in the peripheral blood, making it a predictor of earlier relapse than commonly measured tumor markers (ACE and CA 19-9). In addition, their presence is associated with a significant decrease in recurrence-free survival and overall survival. Studies in colorectal cancer show similar results to those shown for breast cancer: In the retrospective study of Linuma et al, multivariate analysis for relapse-free survival (SSR) and overall survival (SG) found that patients with CTC expression and positive ctDNA had a worse prognosis than the others: SG (hazard ratio [HR], 3.84, 95% CI, 2.41 to 6.22, P .001) and SSR ( HR, 3.02, 95% CI, 1.83 to 5.00, P .001). These results are found in the prospective study by Roder et al, where the detection of CTC in operated patients with colon cancer is associated with 5-year Overall survival (OS)of 68% against 85% in patients without CTC detectable. In multivariate analysis, the results are similar with a significant difference on SG (HR1.94, 95% CI 1.0-3.7, p = 0.04) and SSR (HR 1.94, 95% CI 1.1-3.7, p = 0.044).

E / Determination of microsatellite instability (MSI) status on ctDNA:

Patients with MSI tumors have a better prognosis than microsatellite stability (MSS) patients and have different sensitivities to chemotherapy. The MSI status is currently determined on the operative specimen in pathology by determining the expression of the MLH1-MSH2-MSH6 and PMS2 proteins by immunohistochemistry and by a molecular test determining the instability of microsatellite markers. The determination of the MSI status on the ctDNA is not carried out in current practice but raises several questions: is it systematically detectable on the ctDNA found on peripheral blood when this phenotype is present? Are the ctDNA levels comparable according to the MSI and MSS status?

F / Influence of the surgical technic on the amount of ctDNA:

In order to limit the metastatic spread of CRC, studies have evaluated standard surgical technics, particularly in order to limit the release of ctDNA or CTC.

Studies have compared laparoscopy versus laparotomy on the level of ctDNA and intraoperative CTC in portal and peripheral blood. The results showed a significant decrease in the overall cDNA level in laparoscopic patients. The randomized prospective study of Wind et al reports CTC levels in the laparotomy and laparoscopic groups, respectively 44% vs. 5%. 9% (p = 0.046) in portal blood after mobilization of the tumor. And after resection of the tumor respectively 29% vs. 20% (p = 0.590) in the portal blood. One of the hypothesis of the authors to explain this difference is that laparoscopic tumor mobilization is significantly less important than the one performed during laparotomy.

This hypothesis led to the principle of the "no touch" technic: to achieve the minimum of intraoperative tumor mobilization with an early ligation of mesenteric vessels.

A few low-level studies have compared ADNct and CTC levels in perioperative peripheral blood comparing the "no touch" technic with those that mobilize the tumor first. The results show a tendency to decrease the rates of both markers in the no-touch technic. In the prospective study by Hayashi et al, 8 out of 11 patients (73%) operated according to the "mobilization first" technique had detectable CTCs in portal and postoperative portal blood samples whereas only 1 patient (14%) from the "no touch" group was detected.

G / Objective:

The objective of this work is to compare the amount of ctDNA and CTC in the peripheral blood at D-1, D1 and D3 after colectomy for localized adenocarcinoma using the surgical "no touch" technic against mobilization first and to determine the MSI status on ctDNA.

The standard procedure for hospitalization for patients requiring colectomy for CCR is as follows:

* A preoperative consultation with the surgeon and one with the anesthesiologist.
* Hospitalization the day before the intervention with visit of the surgeon and the anesthesiologist, blood sample of a complete preoperative assessment (D-1).
* Intervention (D0): right or left colectomy depending on tumor localization.
* Systematic blood test after surgery on D1, D3: samples of 4ml tubes for blood count determination, blood Ionogram and assay of C-reactive protein.
* Release on D4 depending on the clinical condition and the results of the blood tests.

As part of the research:

* An information note is given to the subject the day before the intervention and a written statement is collected before the J-1 levy
* During the blood samples taken as part of the treatment, an additional volume is collected 2 samples of 6mL at D-1 then at D1 and D3 to measure the levels of circulating tumor cells and tumor circulating DNA by PCR and the MSI status. There is no blood sample added by the research, the tubes are thus collected at the same time as the standard blood samples of usual perioperative follow-up.

D / ctDNA Extraction, Molecular Tests, and CTC Detection:

The extraction of complementary deoxyribonucleic acid (cDNA) will be performed with an extraction automaton (MaxwellTM) from 6 ml of plasma obtained from the blood sample. The cDNA obtained will be quantified by fluorimetry and quantitative polymerase chain reaction (qPCR). Molecular analyzes will be performed by high-throughput sequencing on targets of interest in colorectal cancer and supplemented with digital PCR targeting mutations previously identified by sequencing the primary tumor (from the operative specimen). A set up of DNA methylation tests can also be done.

Due to the rarity of CTCs, it is necessary to proceed in two steps: i) enrichment followed ii) ScreenCell® detection is a non-invasive technique that allows to enrich from the peripheral blood a cell fraction containing circulating cells The ScreenCell® Molecular Biology (MB) kit then makes it possible to carry out molecular analyzes such as PCRs in order to sequence the gene of interest. This ScreenCell® MB kit allows DNAse free filtration. Before filtration, 6 ml of blood are diluted in 1 ml of the buffer provided. Two minutes after 1.6 ml of the culture medium adapted to the blood cells studied. After filtration, the kit allows extraction of RNA directly from isolated cells in the filter. An adequate volume of the lysis buffer is added directly to the filter capsule (closed in an eppendorf) to extract RNA from the isolated cells in the filter. After centrifugation, the genetic material will be analyzed. For this, a reverse transcriptase will be performed in order to obtain the cDNA of interest.

Statistical analyzes will be performed to compare tumor cell and circulating DNA levels according to non parametric Fisher or chi² tests. A value of p <0.005 is considered significant.

ELIGIBILITY:
Inclusion Criteria:

* men and women, aged over18 years old and more
* colectomy for localized colon adenocarcinoma
* Adenocarcinoma of the colon stage 1,2,3
* Patient having signed the consent

Exclusion Criteria:

* carcinomatosis
* metastatic tumor
* pregnancy and breast feeding

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients, aged over 18 years old and more, undergoing colectomy for non-metastatic adenocarcinoma (stage I, II, III) in the colorectal surgery department at St Antoine Hospital from 01/01/2018 to 1/07/2019 are included in the study. Written consent is obtained at the time of admission.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2019-02-05 (Actual); Primary Completion 2019-08 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Presence of ctDNA | Day 1
  Evaluate the presence of ctDNA on D1 postoperatively by comparing the two methods of surgery: "no touch" method and first mobilization of the tumor in patients with colon cancer
Presence of ctDNA | Day -1
  Evaluate the presence of ctDNA on D-1 postoperatively by comparing the two methods of surgery: "no touch" method and first mobilization of the tumor in patients with colon cancer
Presence of ctDNA | Day 3
  Evaluate the presence of ctDNA on D3 postoperatively by comparing the two methods of surgery: "no touch" method and first mobilization of the tumor in patients with colon cancer

SECONDARY OUTCOMES:
Presence of CTC | Day -1, Day 1 and Day 3
  Evaluate the presence of CTC at D-1, D1 and D3 in peripheral blood by comparing the two methods of surgery between the "no touch" method and first mobilization of the tumor in patients with colon cancer.
MSI status | Day -1, Day 1 and Day 3
  Determine the MSI status on ctDNA in the postoperative period.

CONTACTS AND LOCATIONS:
Overall Officials: Yann Parc, PU-PH, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Department of Digestive Surgery, Hôpital Saint-Antoine, Paris, France